CLINICAL TRIAL: NCT04337957
Title: Elderly Patients With Renal Insufficiency: Reasons for Using the Geriatrician, Modalities and Results of the Geriatric Evaluation, Becoming at One Year
Acronym: NephroG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2019/VA-1
Record Dates: First submitted 2019-07-01; First posted 2020-04-08 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Secondary Evaluation Criteria; Comorbidities and Coexisting Conditions; Motility Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: geriatric nephrology — Collection of the geriatrician's opinion

SUMMARY:
The incidence and prevalence of kidney failure increases with age. Elderly people with chronic kidney disease may have factors of fragility (loss of independence, comorbidities, geriatric syndromes) that can complicate the choice and implementation of the nephrological therapeutic project. Joint and early assessment of these patients by a nephrologist and a geriatrician could help to optimize the definition of care objectives and patient pathway.

There is little data on how nephrologists and geriatricians cooperate and on the description of frailties in elderly patients with renal impairment.

In this context, the objective of this study is to describe in a French university hospital the reasons for the use of geriatricians by nephrologists, the modalities of geriatric evaluation and the socio-demographic and medical characteristics (including geriatric syndromes) of very elderly patients with renal insufficiency, and then to become so at one year.

Year of implementation of this research: 2019 based on data from 2017 and 2019. Approximate number of people likely to be included in the research: 100 patients

DETAILED DESCRIPTION:
There is little data on how nephrologists and geriatricians cooperate and on the description of frailties in elderly patients with renal impairment.

In this context, the objective of this study is to describe in a French university hospital the reasons for the use of geriatricians by nephrologists, the modalities of geriatric evaluation and the socio-demographic and medical characteristics (including geriatric syndromes) of very elderly patients with renal insufficiency, and then to become so at one year.

Secondary objectives :

* describe the modalities of the geriatric evaluation
* describe the socio-demographic, medical characteristics (including fragilities and/or geriatric syndromes) of elderly patients with renal insufficiency
* describe how to become one year old.

Origin and nature of the data collected:

- Socio-demographic, medical and geriatric data (see attached document) based on geriatric assessment medical records (reports of external geriatric consultation and/or intervention by the mobile geriatric team).

The approximate duration of the study will be 9 months. This time includes the time required for statistical analysis and writing an article.

ELIGIBILITY:
Inclusion Criteria:

* 75-year-old patient and older
* Renal insufficiency
* Use in 2017 and 2018 of a geriatric evaluation at the Nîmes University Hospital at the request of nephrologists (mobile geriatric team or external geriatric consultation).

Exclusion Criteria:

* Patient under guardianship, curatorship or judicial protection
* Patient under 75-year-old

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: Very old patients with renal insufficiency
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
reason for the nephrologist's recourse for a geriatric assessment with a geriatric team | up to one year
  geriatric syndromes recorded from medical records

SECONDARY OUTCOMES:
geriatric advice for therapeutic project including dialysis option | up to one year
  rate of geriatric advice for therapeutic project including dialysis option listed from medical records
falls recorded from geriatric assessment medical records | up to one year
  number of falls recorded from geriatric assessment medical records
death,assessment from medical records | at one year
  number of death recorded from medical records
dialyses and death recorded from medical records | at one year
  rate of dialyses and death recorded from medical records

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Nîmes, France